CLINICAL TRIAL: NCT03043690
Title: Clinical Efficacy of an Ammonium Succinate-based Dietary Supplement in Women With Menopausal Symptoms: a Pooled Analysis of the Data From Two Randomized, Multicenter, Double-blinded Placebo-controlled Clinical Trials.
Brief Title: A Pooled Analysis of the Data From Two Studies of Ammonium Succinate for Menopausal Symptoms
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Kuznetsova Irina, Senior Research Fellow, I.M. Sechenov First Moscow State Medical University
Other Study IDs: AMSUCC2
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-02

CONDITIONS: Menopause Related Conditions
Keywords: menopause; ammonium succinate
MeSH Terms: interventions — Succinic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ammonium succinate: Patients in main pooled study group received 2 capsules of ammonium succinate-based dietary supplement (one white, 200 mg, and one orange, 200 mg), once a day, in the morning with a meal, for 90 days.
  Interventions: Dietary Supplement: Ammonium succinate
- Placebo: Patients in placebo study group received 2 capsules of ammonium succinate-based dietary supplement (one white, 200 mg, and one orange, 200 mg), once a day, in the morning with a meal, for 90 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ammonium succinate — 2 capsules of ammonium succinate-based dietary supplement (one white, 200 mg, and one orange, 200 mg), once a day, in the morning with a meal, for 90 days.
  Groups: Ammonium succinate
Other: Placebo — 2 capsules of ammonium succinate-based dietary supplement (one white, 200 mg, and one orange, 200 mg), once a day, in the morning with a meal, for 90 days.
  Groups: Placebo

SUMMARY:
This study is a pooled statistical analysis of the data from 2 studies concerning efficacy of ammonium-succinate based dietary supplement. In both studies group 1 took the ammonium-succinate based dietary supplement and the group 2 took placebo.

DETAILED DESCRIPTION:
Both studies were conducted previously and were randomized, double-blind and placebo-controlled. They followed very similar protocols, were of nearly identical design, had common inclusion and exclusion criteria. Both studies achieved statistical significance for ammonium succinate-based dietary supplement on most of pre-specified endpoints of Greene Climacteric Scale symptoms severity reduction at week 12. Nevertheless, some minor variation in the patient population, both within the studies (e.g., between different centres, as well as seasonal variability) and between the studies can be expected.

Naturally occuring estrogen deficiency over the course of the menopausal transition and postmenopause causes hot flushes and other psychosomatic and vasomotor symptoms. Menopausal hormone therapy is a method of choice, however in many cases it is contraindicated or unacceptable for other reasons. Many alternatives exist, generally acting via estrogen receptors (ER). The dietary supplement tested in the aforementioned studies contains ammonium succinate, which does not bind to ER, instead acting by supporting the Krebs cycle. It does not have phytoestrogenic ingredients.

ELIGIBILITY:
Inclusion Criteria:

* vasomotor and psychosomatic complaints
* ability to comply to study protocol
* signed informed consent

Exclusion Criteria:

* cancer (current or prior, based on medical history)
* conditions requiring planned hospitalization in the next 6 months;
* endocrine diseases with abnormal hormonal secretion (hypercorticism, hyperprplactinemia, hypersomatotropism, thyroid disorders et c.);
* any surgeries within 1 year of the screening;
* hormone therapy within 6 months of the screening;
* psychiatric diseases;
* diabetes mellitus;
* taking other supplements or medications that may affect the climacteric syndrome

Ages: 42 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Both studies chosen for pooled analysis recruited women with vasomotor and psychosomatic complaints, in the late phase of the menopausal transition and postmenopause according to the Stages of Reproductive Aging Workshop +10 classification.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
"Heart beating quickly and strongly" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling tense or nervous" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Difficulty in sleeping" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Excitable" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Attacks of panic" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Difficulty in concentrating" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling tired or lacking in energy" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of interest in most things" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling unhappy or depressed" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Crying spells" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Irritability" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling dizzy or faint" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Pressure or tightness in head or body" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Parts of body feeling numb or tingling" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Headaches" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Muscle or joint pains" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of feeling in hands or feet" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Breathing difficulties" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Hot flushes" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Sweating at night" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of interest in sex" symptom (Greene Climacteric Scale) | Week 12
  Statistically significant reduction in designated symptom severity, compared between arms

SECONDARY OUTCOMES:
Spilberger-Hanin (Situational anxiety) | Week 12
  The decrease of situational anxiety, measured as statistically significant reduction of the score in corresponding subscale
Spilberger-Hanin (Personal anxiety) | Week 12
  The decrease of personal anxiety, measured as statistically significant reduction of the score in corresponding subscale
Spilberger-Hanin (Actual anxiety) | Week 12
  The decrease of actual anxiety, measured as statistically significant reduction of the score in corresponding subscale. Actual anxiety as a sum of situational and personal anxiety scores was introduced by Hanin in his modification of original State-Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Irina V Kuznetsova, Principal Investigator — Sechenov First Moscow Medical University
Locations (1):
- Sechenov First Moscow Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radzinskii VE, Kuznetsova IV, Uspenskaya YB, Repina NB, Gusak YK, Zubova OM, Burchakov DI, Osmakova AA. Treatment of climacteric symptoms with an ammonium succinate-based dietary supplement: a randomized, double-blind, placebo-controlled trial. Gynecol Endocrinol. 2016 Oct;32(sup2):64-68. doi: 10.1080/09513590.2016.1232686. PMID 27759458
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. Menopause. 2012 Apr;19(4):387-95. doi: 10.1097/gme.0b013e31824d8f40. PMID 22343510
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 2008 Sep-Oct;61(1-2):78-84. doi: 10.1016/j.maturitas.2008.09.011. PMID 19434881